CLINICAL TRIAL: NCT07021066
Title: A Phase 1 Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M05D1 in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M05D1 in Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BL-M05D1-ST-101
Record Dates: First submitted 2025-05-23; First posted 2025-06-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Gastric Adenocarcinoma; Advanced Pancreatic Ductal Adenocarcinoma; Esophageal Adenocarcinoma; Biliary Tract Cancer; Other Solid Tumors
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental BL-M05D1 administered Day 1 per cycle (Experimental): BL-M05D1 will be administered on Day 1 by intravenous (IV) infusion every 3 weeks
  Interventions: Drug: BL-M05D1

INTERVENTIONS:
Drug: BL-M05D1 — BL-M05D1 will be administered on D1 every 3 weeks.

SUMMARY:
The objective of this study is to evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M05D1 in Subjects with Advanced or Metastatic Solid Tumors.

DETAILED DESCRIPTION:
This is a multicenter Phase 1, open-label study to evaluate the safety, tolerability, pharmacokinetic profile, and initial efficacy of BL-M05D1 in subjects with unresectable locally advanced or metastatic solid tumors that are known to potentially express CLDN18.2 as defined below that have recurred or progressed on at least 1 line of prior systemic therapy (including adjuvant/neoadjuvant), have no other standard of care options, and have no available curative options.

This study will be conducted in three parts (dose escalation, dose finding and dose expansion). Subjects will be dosed on Day 1 on a continuous 21-day treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form voluntarily and agreed to follow the program requirements
2. Age: ≥18 years
3. Has a life expectancy of ≥3 months
4. Has documented locally advanced or metastatic solid tumor(s) that are known to potentially express CLDN18.2 as defined below that have recurred or progressed on at least 1 line of prior systemic therapy (including adjuvant/neoadjuvant), have no other standard of care options, and have no available curative options, including:

   1. Gastric or gastroesophageal junction (G/GEJ) adenocarcinoma (AC): Subjects with CLDN18.2, human epidermal growth factor receptor 2 (HER2), PD-L1 and/or microsatellite instability high (MSI-H)/ mismatch repair deficiency (dMMR) positive tumors must have received targeted treatment in their prior lines of therapy.
   2. Pancreatic ductal AC (PDAC): Subjects may enter screening prior to completing the first line of standard therapy.
   3. Esophageal AC (EAC): Subjects with HER2, PD-L1 and/or MSI-H/dMMR positive tumors must have received targeted treatment in their prior lines of therapy.
   4. Biliary tract cancers (BTCs): Subjects with HER2 overexpression, NTRK fusions, KRAS mutations, IDH1 mutations, FGFR2 fusions, BRAF mutations and/or MSI-H/dMMR positive tumors must have received targeted treatment in their prior lines of therapy.
   5. Other solid tumors not specified above may be included IF they have documented CLDN18.2 expression by IHC (1+). As applicable per standard of care, subjects with HER2 and/or PD-L1 positive tumors must have received targeted treatment in their prior lines of therapy, and subjects with MSI-H or dMMR positive tumors must have received immune checkpoint inhibitor.
5. Agree to provide most recent existing tumor samples (formalin-fixed paraffin-embedded [FFPE] tissue block or slides) from primary or metastatic sites (see details in Section 7.1.1) for tissue-based evaluation of CLDN18.2 expression. A fresh biopsy is required if no archival/FFPE block or slides are available. Re-biopsy is recommended if the subject previously received a CLDN18.2-directed treatment.
6. Has at least one measurable lesion based on RECIST (Response Evaluation Criteria in Solid Tumors) v1.1
7. Has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1
8. Toxicity of previous antitumor therapy has returned to Grade ≤1 as defined by the National Cancer Institute (NCI) CTCAE v5.0, except for alopecia and endocrinopathies controlled by replacement therapy that must be Grade ≤2
9. Has no serious cardiac dysfunction, left ventricular ejection fraction ≥50%
10. Has adequate organ function before enrollment, defined as:

    1. Marrow function: Absolute neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥100×109/L, hemoglobin (Hb) ≥9.0 g/dL (blood transfusion, platelet transfusion, erythropoietin, hematopoiesis agents, and granulocyte-colony stimulating factor [G-CSF] use are not allowed 1 week prior to screening)
    2. Hepatic function: Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) (≤3×ULN for subjects with Gilbert's syndrome or liver metastasis at baseline), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) without liver metastasis ≤3.0×ULN, AST and ALT with liver metastasis ≤5.0×ULN NOTE: For patients with Gilbert's syndrome, conjugated bilirubin ≤1.5×ULN and TBIL <3.0×ULN in the absence of liver metastases.
    3. Renal function: Creatinine (Cr) clearance ≥60 mL/min (Cockcroft-Gault equation) or estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73 m2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation)
11. Coagulation parameters: International normalized ratio (INR) ≤1.5×ULN, and activated partial thromboplastin time (aPTT) ≤1.5×ULN, unless receiving anticoagulation therapy with prothrombin time and aPTT levels within the intended therapeutic range
12. Urine protein ≤2+ or ≤1000 mg/24 hours
13. Sexually active fertile subjects and their partners must agree to use highly effective methods of contraception (defined in Appendix E) during the course of the study and after the last dose of study treatment (7 months for women and 4 months for men). An additional contraceptive method, such as a barrier method (eg, condom), is recommended.
14. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and must be nonlactating. Female subjects are considered WOCBP unless one of the following criteria are met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman >45 years old in the absence of other biological or physiological causes. In addition, females <55 years old must have a serum follicle stimulating hormone (FSH) level >40 mIU/mL to confirm menopause.

Note: Documentation may include review of medical records, medical examination, or medical history interview by study site staff.

Exclusion Criteria:

1. Chemotherapy, biological therapy, immunotherapy, radical radiotherapy, targeted therapy (including small molecule inhibitor of tyrosine kinase), and other antitumor therapy within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration; major surgery within 4 weeks prior to the first administration; mitomycin and nitrosoureas treatment within 6 weeks prior to the first administration
2. Subjects with history of severe heart disease, such as symptomatic congestive heart failure (CHF) ≥ Grade 2 (CTCAE v5.0), New York Heart Association (NYHA) ≥ Grade 2 heart failure at any time, or history of myocardial infarction or unstable angina pectoris within 6 months before enrollment
3. Subjects with prolonged QT interval corrected ([QTcF] >470 msec), complete left bundle branch block, Grade 3 atrioventricular block
4. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc. Subjects with well-controlled type 1 diabetes, hypothyroidism, and skin diseases that do not require systemic treatment (such as vitiligo, psoriasis) are permitted. For autoimmune conditions that are active but stable and low grade on systemic therapy, discussion with the medical monitor is required prior to screening
5. Subjects with other prior malignancies except for: basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or carcinoma in situ after adequate resection, or other malignancy treated with curative intent with a disease-free interval of at least 3 years prior to screening
6. Subjects with poorly controlled hypertension by two types of antihypertensive drugs (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg)
7. Subjects with advanced or clinically significant lung diseases, such as poorly controlled chronic obstructive pulmonary disease and asthma, restrictive lung disease, pulmonary hypertension, etc.
8. Subjects who have a history of noninfectious interstitial lung disease (ILD)/ pneumonitis that required treatment with steroids, have current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening
9. Subjects with stroke or transient ischemic attack (TIA) within 6 months before enrollment
10. Subjects with a thromboembolic event (eg, deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 6 months before enrollment except for those who are clinically stable and receiving treatment with adequate anticoagulant therapy for at least 3 weeks before enrollment
11. Subjects with primary tumors in the central nervous system (CNS) and active or untreated CNS metastases and/or carcinomatous meningitis should be excluded. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and no requirements for corticosteroids 14 days prior to dosing with the investigational product (IP). Patients on low dose corticosteroids (<20 mg prednisone or equivalent/day) may participate.
12. Subjects with pre-existing Grade ≥2 peripheral neuropathy
13. Subjects who have a history of anaphylaxis or severe hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies or any of the components of BL-M05D1
14. Subjects who are receiving treatment with systemic glucocorticoids >10 mg/day equivalent of prednisone, except for the treatment of chronic obstructive pulmonary disease, antiemetic, infusion reactions; however, treatment with low dose glucocorticoids (≤10 mg/day equivalent of prednisone) is permitted. The chronic use of topical, inhaled, and locally injected steroids is permitted
15. Subjects who have received treatment with anthracyclines with a cumulative dose exceeding 360 mg/m2
16. Subjects with known human immunodeficiency virus (HIV) infection (HIV antibody positive). Subjects are allowed to participate if all the following criteria are met:

    1. Undetectable HIV RNA and CD4 count ≥ 350 cells/μL at screening;
    2. No AIDS-defining opportunistic infection within 12 months prior to screening;
    3. On stable antiretroviral therapy (ART) for at least 4 weeks prior to enrollment with projected continuation of ART as clinically indicated while on the study.
17. Subjects with known active hepatitis B virus (HBV) infection (positive HBsAg test). Subjects with a chronic inactive HBV infection are eligible if all the following criteria are met:

    1. Have an HBV DNA viral load < 500 IU/mL;
    2. Have normal AST and ALT, OR if liver metastasis is present, have AST and ALT <3×ULN which are not attributed to HBV infection;
    3. Are on antiviral treatment, as clinically indicated.
18. Subjects with known active hepatitis C virus (HCV) infection (HCV antibody positive and HCV-RNA > the lower limit of detection). Subjects with a positive anti-HCV antibody are eligible only if quantitative polymerase chain reaction (PCR) is negative for HCV RNA
19. Subjects with known active tuberculosis
20. Subjects with active infections requiring IV antibiotic, antiviral, or antifungal treatment, such as severe pneumonia, bacteremia, sepsis, etc., within 1 week prior to first dose of study treatment. Subjects on stable oral antimicrobials with no clinical or laboratory evidence of active infection are eligible
21. Subjects who are pregnant, breastfeeding, or planning to become pregnant during the study
22. Other conditions that the investigator believes are not suitable for participating in this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Participants with Dose-limiting toxicities | 1 year
  A DLT is defined as the following:
  Toxicity that results in a >14-day delay in treatment
  - Hematologic toxicities
  Grade 4 neutrophil count decreased lasting >7 days
  Grade ≥3 febrile neutropenia of any duration
  Grade ≥3 platelet count decreased with clinically significant hemorrhage
  Grade 4 thrombocytopenia lasting >72 hours
  - Nonhematologic toxicities
  Death not clearly related to disease progression or extraneous cause
  Hy's law cases
  Grade ≥3 nonhematologic toxicities, except for:
  Grade 3 nausea/vomiting or diarrhea for less than 72 hours with adequate antiemetic and other supportive care
  Grade 3 fatigue for less than 1 week
  Grade ≥3 electrolyte abnormality that lasts up to 72 hours, is not clinically complicated, and resolves spontaneously or responds to conventional medical interventions
  Grade ≥3 amylase or lipase that is not associated with symptoms or clinical manifestations of pancreatitis
Participants with Serious Adverse Events (SAEs) and treatment-emergent adverse events (TEAEs) | 1 year
  Measuring the number of patients with serious adverse events (SAEs) and treatment-emergent adverse events (TEAEs)
Participants with abnormal physical examination findings | 1 year
  Measure the number of participants with abnormal physical examination findings.
Participants with ability to care for themselves, daily activity, and physical activity | 1 year
  Measure the change in participants with Eastern Clinical Oncology Group (ECOG) Scale of Performance Status. The scale is 0-4 with 0 being the fully active (best outcome) and 4 being completely disabled (worst outcome)
Participants with abnormal ECG and ECHO/MUGA reading | 1 year
  Patients with abnormal ECG parameters (including the change from-baseline ECG parameters: heart rate [HR]; PR; QTcF; and QRS intervals [∆HR, ∆PR, ∆QTcF, and ∆QRS]), and ECHO/MUGA findings
Participants with abnormal lab results | 1 year
  Measure the number of participants with abnormal clinical laboratory values
To determine the maximum tolerated dose (MTD) if reached or maximum administered dose (MAD) and two or more recommended doses for expansion (RDEs) of BL-M05D1 in metastatic or unresectable tumors | 1 year
  The actual number of subjects enrolled and dose levels to be explored in this study will depend on the MTD and/or RDE based on DLTs reported during the DLT observation period.

SECONDARY OUTCOMES:
Cmax of BL-M05D1 | 1 year
  Calculate maximum (peak) observed concentration of BL-M05D1
Cmax of anti-BL-M05D1 antibodies | 1 year
  Calculate maximum (peak) observed concentration of anti-BL-M05D1 antibodies
Cmax of free payload ED-04 | 1 year
  Calculate maximum (peak) observed concentration of free payload ED-04
Tmax of BL-M05D1 | 1 year
  Calculate time of maximum observed concentration of BL-M05D1
Tmax of anti-BL-M05D1 antibodies | 1 year
  Calculate time of maximum observed concentration of anti-BL-M05D1 antibodies
Tmax of free payload ED-04 | 1 year
  Calculate time of maximum observed concentration of free payload ED-04
AUC(0-8) of BL-M05D1 | 1 year
  Calculate area under the serum concentration-time curve of BL-M05D1 from time 0 to 8 hours
AUC(0-8) of anti-BL-M05D1 antibodies | 1 year
  Calculate area under the serum concentration-time curve of anti-BL-M05D1 antibodies from time 0 to 8 hours
AUC(0-8) of free payload ED-04 | 1 year
  Calculate area under the serum concentration-time curve of free payload ED-04 from time 0 to 8 hours
AUC(last) of BL-M05D1 | 1 year
  Calculate area under the serum concentration-time curve up of BL-M05D1 to the last quantifiable time0 to 8 hours
AUC(last) of anti-BL-M05D1 antibodies | 1 year
  Calculate area under the serum concentration-time curve up of anti-BL-M05D1 antibodies to the last quantifiable time0 to 8 hours
AUC(last) of free payload ED-04 | 1 year
  Calculate area under the serum concentration-time curve up of free payload ED-04 to the last quantifiable time
Overall Response Rate (ORR) | 1 year
  To assess the clinical efficacy of BL-M05D1 as measured by ORR using RECIST criteria v 1.1
Disease Control Rate (DCR) | 1 year
  To assess the clinical efficacy of BL-M05D1 as measured by DCR using RECIST criteria v 1.1
Time To Response (TTR) | 1 year
  To assess the clinical efficacy of BL-M05D1 as measured by TTR using RECIST criteria v 1.1
Progression-Free Survival (PFS) | 1 year
  To assess the clinical efficacy of BL-M05D1 as measured by PFS using RECIST criteria v 1.1
Overall Survival (OS) | 1 year
  To assess the clinical efficacy of BL-M05D1 as measured by OS using RECIST criteria v 1.1
Duration of response (DoR) | 1 year
  To assess the clinical efficacy of BL-M05D1 as measured by DoR using RECIST criteria v 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tannenbaum, Study Director — SystImmune Inc.
Locations (17):
- United States (17):
  - Mayo Clinic Cancer Center- Phoenix, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - University of Colorado Health, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute - Oncology Partners, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - NEXT Oncology- Austin, Austin, Texas
  - NEXT Oncology- Dallas, Dallas, Texas
  - MD Anderson, Houston, Texas
  - NEXT Oncology San Antonio, San Antonio, Texas
  - START Center for Care Center- San Antonio, San Antonio, Texas
  - Baylor Scott and White Medical Center- Temple Clinic, Temple, Texas

IPD SHARING:
Plan to Share IPD: No